CLINICAL TRIAL: NCT05881772
Title: Acute Effect of Photobiomodulation Therapy on Quadriceps Muscle Strength in Patients With Chronic Kidney Failure on Hemodialysis: a Crossover Randomized Clinical Trial
Brief Title: Acute Effect of Photobiomodulation on Quadriceps Muscle Strength in Patients With Chronic Kidney Failure on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Jociane Schardong, Doctor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Laser_HD
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Renal Insufficiency, Chronic; Renal Dialysis
Keywords: Low-Level Light Therapy; Renal Insufficiency, Chronic; Randomized Controlled Trial
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1 (Active Comparator): It will be applied a dose of 30J (180J per leg) of laser radiation through a cluster with four diodes, wavelength of 830 nm and power of 800mW (200mW/diode), HTM® (model Fluence Maxx, São Paulo, Brazil) on quadriceps muscle.
  Interventions: Other: Photobiomodulation
- Experimental 2 (Active Comparator): It will be applied a dose of 60J (360J per leg) of laser radiation through a cluster with four diodes, wavelength of 830 nm and power of 800mW (200mW/diode), HTM® (model Fluence Maxx, São Paulo, Brazil) on quadriceps muscle.
  Interventions: Other: Photobiomodulation
- Experimental 3 (Active Comparator): It will be applied a dose of 90J (540J per leg) of laser radiation through a cluster with four diodes, wavelength of 830 nm and power of 800mW (200mW/diode), HTM® (model Fluence Maxx, São Paulo, Brazil) on quadriceps muscle.
  Interventions: Other: Photobiomodulation
- Placebo group (Placebo Comparator): The placebo treatment will be performed with the equipment HTM® (model Fluence Maxx, São Paulo, Brazil) turned off.
  Interventions: Other: Photobiomodulation

INTERVENTIONS:
Other: Photobiomodulation — It will be applied a dose of laser radiation through a cluster with four diodes, wavelength of 830 nm and power of 800mW (200mW/diode), HTM® (model Fluence MAXX, São Paulo, Brazil). For application, the patient will be positioned in a sitting position and the treatment will be performed with the fixed probe in contact with the skin at an angle of 90º, using the continuous emission mode. The therapy will be applied to the quadriceps muscle, bilaterally.
  Other Names: Low level laser therapy

SUMMARY:
Chronic kidney disease (CKD) consists of kidney damage and progressive and irreversible loss of kidney function. The aim of this study is to evaluate the acute effect of different doses of photobiomodulation therapy on quadriceps isometric muscle strength, pain and muscle fatigue of lower limbs and to establish the ideal dose for patients with CKD on hemodialysis. Patients will be submitted to application of photobiomodulation therapy in the quadriceps muscle. Immediately after, the maximum isometric strength test of the quadriceps will be performed.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) consists of kidney damage and progressive and irreversible loss of kidney function. In the most advanced stage of the disease the patients require hemodialysis (HD) and present alterations such as: sarcopenia, cardiovascular disorders, increased systemic inflammation, muscle weakness and fatigue. These factors negatively affect the individual's functionality, impacting the increase in hospitalization and mortality rates. Photobiomodulation (FBM) has shown positive results in different populations on improving performance during exercise, reducing fatigue and markers of muscle damage. The aim of this study is to evaluate the acute effect of FBM therapy on quadriceps muscle strength, pain and muscle fatigue in patients with CKD on HD and to establish the ideal therapeutic dose. Patients will be submitted to application of four applications with different doses of FBM (30J, 60J, 90J and placebo) in the quadriceps muscle, in random order and one week interval between them for washout. Patients and evaluators will be blinded to the intervention protocol. The following assessments will be performed prior to FBM: subjective perception of exertion (by modified Borg scale), muscle fatigue (by analysis of blood lactate) and pain perception (by numeric pain scale). After the FBM application, the maximum isometric strength test of the quadriceps will be performed by dynamometry. Immediately after performing the strength test, all assessments will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD on HD for a period ≥ 3 months;
* Age between 18-80 years old;
* Patients of both sexes;
* Dialysis with a weekly frequency of 3 times/week;
* Adequate urea clearance rate (Kt/V ≥ 1.2 or URR ≥65%).

Exclusion Criteria:

* Cognitive dysfunction that prevents the performance of the assessments, as well as inability to understand and sign the informed consent form;
* Epidermal lesions at the site of application of photobiomodulation therapy;
* Patients with recent stroke sequelae (three months);
* Recent acute myocardial infarction (two months);
* Uncontrolled hypertension (SBP>230 mmHg and DBP>120 mmHg);
* HF grade IV according to the New York Heart Association or decompensated;
* Unstable angina;
* Peripheral vascular changes in lower limbs such as deep venous thrombosis;
* Disabling osteoarticular or musculoskeletal disease;
* Uncontrolled diabetes (blood glucose > 300mg/dL);
* Febrile state and/or infectious disease;
* Systemic lupus erythematosus;
* Patients undergoing cancer treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Maximal isometric muscle strength of the quadriceps | Immediately after the aplication of photobiomodulation therapy.
  Maximal isometric muscle strength of the quadriceps will be assessed by dynamometry.

SECONDARY OUTCOMES:
Muscle pain of lower limbs | Baseline and immediately after the dynamometry.
  Muscle pain of lower limbs will be assessed by the numeric pain scale (NPS). Zero means no pain and 10 maximum pain.
Fatigue | Baseline and immediately after the dynamometry.
  Fatigue of lower limbs by the modified Borg subjective perceived exertion scale Modified Borg (Borg Scale). Zero means no effort or fatigue and 10 maximum effort or fatigue.
Fatigue | Baseline, immediately after dynamometry, at 3 and 6 minutes.
  Fatigue of lower limbs by blood lactate dosage.

CONTACTS AND LOCATIONS:
Overall Officials: Jociane Schardong, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No